CLINICAL TRIAL: NCT01049854
Title: CD34+Stem Cell Selection for Patients Receiving Partially Matched Family or Matched Unrelated Adult Donor Allogeneic Stem Cell Transplantations for Malignant and Non-Malignant Disease
Brief Title: CD34+Selection for Partially Matched Family or Matched Unrelated Adult Donor Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York Medical College (Other)
Responsible Party: Principal Investigator, Mitchell Cairo, Principal Investigator, New York Medical College
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L 10,321; NYMC 525 (Other: NYMC)
Record Dates: First submitted 2008-05-05; First posted 2010-01-15 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Leukemia; Lymphoma; Bone Marrow Failure; Immunodeficiencies; Histiocytosis; Sickle Cell Disease; Beta Thalassemia; Inborn Errors of Metabolism
Keywords: unrelated donor transplant; CD34 selection
MeSH Terms: conditions — Leukemia; Lymphoma; Bone Marrow Failure Disorders; Immunologic Deficiency Syndromes; Histiocytosis; Anemia, Sickle Cell; beta-Thalassemia; Metabolism, Inborn Errors | interventions — Whole-Body Irradiation; Thiotepa; Cyclophosphamide; Antilymphocyte Serum; Busulfan; Melphalan; fludarabine phosphate; Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Thiotepa/Cyclophosphamide/ATG (Experimental): Full intensity with TBI
  Interventions: Drug: Full Intensity with TBI
- Busulfan/Melphalan/ATG (Experimental): Full intensity without TBI
  Interventions: Drug: Full Intensity
- Busulfan/Fludarabine/Alemtuzumab (Experimental): Reduced Intensity Chemotherapy
  Interventions: Drug: Reduced Intensity
- Fludarabine/Cyclophosphamide/ATG (Experimental): Reduced Intensity Chemotherapy for Fanconi Anemia
  Interventions: Drug: Reduced Intensity (Fanconi)

INTERVENTIONS:
Drug: Full Intensity with TBI — Patients will start their pre-conditioning regimen on Day -8. Fractionated TBI will be administered twice daily for 3 days on Days -8, -7, and -6. Patients will receive Thiotepa on Days -5, -4, Cyclophosphamide on Days -3, -2 and rabbit antithymocyte globulin on Days -4, -3, -2 and -1. The stem cell infusion will be performed on Day 0. GM-CSF hematopoietic growth factor will start on Day 0. GVHD prophylaxis will consist of tacrolimus only.
  Other Names: ThioTepa; Cytoxan; Atgam
  Arms: Thiotepa/Cyclophosphamide/ATG
Drug: Full Intensity — Patients will start their pre-conditioning regimen on Day -9. Patients will receive busulfan twice daily on Days - 8, -7, -6, and -5 and Melphalan on Days -4, -3 and -2 and rabbit antithymocyte globulin on Days -4, -3, -2 and -1 with stem cell infusion on Day 0. GM-CSF hematopoietic growth factor will start on Day 0. GVHD prophylaxis will consist of tacrolimus only.
  Other Names: Myleran; Alkeran; Atgam
  Arms: Busulfan/Melphalan/ATG
Drug: Reduced Intensity — Patients will start their GVHD prophylaxis with Tacrolimus on Day -9. Patients will receive busulfan twice daily on Days -8, -7, -6, and -5; fludarabine on Days -7, -6, -5, -4, -3 and -2 and alemtuzumab on Days -5, -4, -3, -2, and -1. The stem cell infusion will be performed on Day 0. GVHD prophylaxis will consist of tacrolimus only.
  Other Names: Fludara; Myleran; Campath
  Arms: Busulfan/Fludarabine/Alemtuzumab
Drug: Reduced Intensity (Fanconi) — Patients will start their pre-conditioning regimen on Day -6. Patients will receive TBI as a single fraction on Day -6. Patients will receive fludarabine and cyclophosphamide on Days - 5, -4, -3, and -2 and antithymocyte globulin (horse) on Days -5, -4, -3, -2 and -1. The stem cell infusion will be performed on Day 0. GVHD prophylaxis will consist of tacrolimus only.
  Other Names: Fludara; Cytoxan; Atgam
  Arms: Fludarabine/Cyclophosphamide/ATG

SUMMARY:
CD34+ stem cell selection in children, adolescents and young adults receiving partially matched family donor or matched unrelated adult donor allogeneic bone marrow or peripheral blood stem cell transplant will be safe and well tolerated and be associated with a low incidence of serious (Grade III/IV) acute and chronic graft versus host disease (GVHD).

DETAILED DESCRIPTION:
The selection of CD34+ cells is associated with the simultaneous depletion of T cells that are responsible for severe acute and chronic graft versus host disease (GVHD). Successful engraftment is reported in adult patients with malignant and non-malignant disease who received CD34+ selected stem cells from HLA-matched or mismatched mobilized peripheral blood (PBSC) or bone marrow.

Study Design:

Selected patients defined in the eligibility criteria will enrolled on this study. Patients will receive one of either full intensity or reduced intensity regimen based on the patient's disease status, organ function and performance and determined by the PI and will have peripheral blood undergo CD34 selection.

ELIGIBILITY:
Inclusion Criteria:

* Adequate renal function defined as:Serum creatinine <1.5 x normal, or Creatinine clearance or radioisotope GFR >60 ml/min/m2 or an equivalent GFR as determined by the institutional normal range.
* Adequate liver function defined as:Total bilirubin <1.5 x normal, or SGOT (AST) or SGPT (ALT) <3.0 x normal
* Adequate cardiac function defined as:Shortening fraction >27% by echocardiogram, or Ejection fraction of >47% by radionucleotide angiogram or echocardiogram.
* Adequate pulmonary function defined as:Uncorrected DLCO >50% by pulmonary function test. For children who are uncooperative, no evidence of dyspnea at rest, no exercise intolerance, and a pulse oximetry >94% on room air.

Eligibility for Reduced Intensity Regimen:

* Adequate renal function defined as:Serum creatinine 2.0 x normal, or creatinine clearance or radioisotope GFR > 40 ml/min/m2 or an equivalent GFR as determined by the institutional normal range.
* Adequate liver function defined as:Total bilirubin < 2.5 x normal; or SGOT (AST) or SGPT (ALT) < 5.0 x normal.
* Adequate cardiac function defined as:Shortening fraction of >25% by echocardiogram, or Ejection fraction of >40% by radionuclide angiogram or echocardiogram.
* Adequate pulmonary function defined as:DLCO >35% by pulmonary function test. For children who are uncooperative, no evidence of dyspnea at rest, no exercise intolerance, and a pulse oximetry >94% in room air.

Exclusion Criteria:

* Pregnancy/Breast Feeding: Females who are pregnant or breast-feeding are not eligible.
* Infection: Patients with documented uncontrolled infection at the time of study entry are not eligible.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-09; Primary Completion 2017-11 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
The safety CD34+ stem cell selection | 100 days
  serious adverse events will be monitored post transplant to determine if there is an increase vs. historical data related to the CD34+ selection

SECONDARY OUTCOMES:
Immune reconstitution (T, B, DC) following CD34+ selection | 3 years
  immune subsets will be drawn post transplant to determine the rate of reconstitution post CD34+ transplant to determine if this process increases or decreases the reconstitution time.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell S Cairo, MD, Principal Investigator — New York Medical College
Locations (1):
- New York Medical College, Valhalla, New York, United States